CLINICAL TRIAL: NCT05087225
Title: Suspicion of Hypoglycemic Effect of mRNA Based Vaccines (Polyethylene Glycol) Will Happen , Observational Study at Saudia Arabia
Brief Title: Suspicion of Hypoglycemic Effect of mRNA Based Covid-19 Vaccines (Polyethylene Glycol) Will Happen , Observational Study on Diabetic Patients at Saudia Arabia
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Ministry of Health, Saudi Arabia (Other Government)
Responsible Party: Principal Investigator, Amr kamel khalil Ahmed, Ministry of health , saudia arabia, Ministry of Health, Saudi Arabia
Other Study IDs: ministry of health saudia
Record Dates: First submitted 2021-10-20; First posted 2021-10-21 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Diabetic Complication; Covid19 Virus Infection; Hypoglycemia; Polyethylene Glycol Adverse Reaction
MeSH Terms: conditions — Diabetes Complications; COVID-19; Hypoglycemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: polyethelyene glycol — the excipients at covid-19 vaccines

SUMMARY:
vaccines for covid-19 are gold strategy and great achievement at this century for protection against complications of covid-19 , development of many vaccines with different technology represent a big challenge for this disease so the world live bad days and the vaccines save world to see the light once again , mRNA based vaccines have a new technology which designed before for cancer therapy, this technology is very effective , producible and fast for future disease targets but these vaccine must contain excipients for preservation of this technology mRNA so we now study these side effects of excipients and we suspect that polyethylene glycol as excipients have big role at hypoglycemic effects with antidiabetic medications like metformin and insulin especially at children and older age

DETAILED DESCRIPTION:
diabetics patients as chronic diseases represent high percentage at all the world and high priority for vaccines against covid-19 so we will focus on these group as need more attention and need best health and quality of life so my study concentrate on diabetics patients from 12 years to 80 years who were taken mRNA based vaccines and suffer from recurrent hypoglycemia , i will check the blood glucose one month after the first or second injection of mRNA based vaccines Pfizer or moderna vaccines and study all medicines taken by patients and suspect what's happen is there is hypoglycemic effect or nor by following up the readings of blood glucose by glucometers or CGM

there are previous studies about relation of metformin and polyethylene glycol injection and this study conclude that The subcutaneous injection of PEX168 once a week can effectively, continuously and safely improve HbA1c levels in patients with T2D when combined with metformin ( Gao F, Lv X, Mo Z, Ma J, Zhang Q, Yang G, Liu W, Li Q, Zhou J, Bao Y, Jia W. Efficacy and safety of polyethylene glycol loxenatide as add-on to metformin in patients with type 2 diabetes: A multicentre, randomized, double-blind, placebo-controlled, phase 3b trial. Diabetes Obes Metab. 2020 Dec;22(12):2375-2383. doi: 10.1111/dom.14163. Epub 2020 Sep 6. PMID: 32744358.

ELIGIBILITY:
Inclusion Criteria:

- Male and female subjects between the ages of 12 and 80 years, inclusive, with Type 1 or 2 diabetes mellitus as defined by the American Diabetes Association (Diabetes care, Vol. 21: S5- S19, 1998) for more than one year.

Exclusion Criteria:

* under 12 years above 80 years undergone bariatric surgery no exercises during testing

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population is a group of individuals selected on the basis of inclusion and exclusion criteria which relate to the variables being studied. It is the population from which the sample population will be randomly or purposively selected
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-11-11 (Estimated); Primary Completion 2022-03-11 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
hypoglycemic effects of polyethylene glycol as excipients covid-19 vaccines at diabetic patients | 6 month
measurement of blood glucose one month after first or second shot of mRNA based covid-19 vaccines | 6 month

SECONDARY OUTCOMES:
enhancements of hypoglycemic effects of metformin and insulin by PEG | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- ministry of health , First health cluster , Riaydh, Riyadh, N/A (Non-US), Saudi Arabia

IPD SHARING:
Plan to Share IPD: No